CLINICAL TRIAL: NCT04810468
Title: Study of Malnutrition inPrimary School Children in Tema City, Sohag Governorate, Egypt to Evaluate the Most Significant Factors Affecting it.
Brief Title: Study of Malnutrition in Primary School Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Naeem Basta, Resident doctor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-21-03-02
Record Dates: First submitted 2021-03-14; First posted 2021-03-23 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Malnutrition, Child
Keywords: Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: The study asses the prevelance malnutrition in primary school children by using anthropometric measurment and asses the sociodemographic data and hygiene information and dietary habits affecting it
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children in primary school (Other): anthropometric measurment will take from each participiant in study to asses wheight ,height ,BMl and also use aquestionnaire yo asses the Sociodemographic data,dietary habits ,hygiene information
  Interventions: Other: Anthropometric measurment

INTERVENTIONS:
Other: Anthropometric measurment — Anthropometric measurment used to asses the wheight in kelogram and asses height in cetemeter and also asses BMI

SUMMARY:
Study of malnutrition in primary school age children aim to asses the prevelance of malnutrition amoung the children in this age group and also ldintified the factors that affect in malnutrition between the children and the study will done in two primary school one present in rural area and another in urban area to compare the factor and the result that affect in both two different area

DETAILED DESCRIPTION:
Study of malnutrition in primary school age children aim to asses the prevelance of malnutrition amoung the children in this age group and also ldintified the factors that affect in malnutrition between the children and the study will done in two primary school one present in rural area and another in urban area to compare the factor and the result that affect in both two different area investigators in this study will use anthropometric measurment to asses wheight and height and BMI and also collect sociodemographic data from participant for Ex father and mother education and age ,sex,place of residence,father and mother jop, mean income.

and also collect data about hygine lnformation for Ex safe and cleen drink water , presence of toilet ,wash hand before and after eating and cooking ,clean nail .

Other data will be collected from participant about dietary habits for Ex how many times eating meat, paultary ,fish in week and how many times eating vegetable,fruits ege milk in day .

This all data will be analysed by use the proper statical analysis system and finally the results will obtained

ELIGIBILITY:
Inclusion Criteria:

* healthy Children who agree the participate in study (6-12) years old .
* Both sexes.

Exclusion Criteria:

* Children below sex years or above 12 years .
* children not in primary school .
* children who refuse participate in study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2021-03-20 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Height measure for the all participant | Measuring the height will take one month
  Height measure for the all participant in cm
Weight measure for the all participant | Weight measure for the all participant will take one month
  Weight measure for the all participant in kg
Sociodemographic data collection | One week
  Sociodemographic data include father and mother education ,age , sex,mean out come, father and mother job,place of residence
Dietary habits data collection | One week
  Dietary habits as how many time eating meat ,fish , vegetable Fruits and another health food

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Abdel Wahed WY, Hassan SK, Eldessouki R. Malnutrition and Its Associated Factors among Rural School Children in Fayoum Governorate, Egypt. J Environ Public Health. 2017;2017:4783791. doi: 10.1155/2017/4783791. Epub 2017 Oct 23. PMID 29201063
- [Background] de Onis M, Blossner M, Borghi E. Prevalence and trends of stunting among pre-school children, 1990-2020. Public Health Nutr. 2012 Jan;15(1):142-8. doi: 10.1017/S1368980011001315. Epub 2011 Jul 14. PMID 21752311